CLINICAL TRIAL: NCT00002149
Title: Acupuncture and Herbal Treatment of Chronic HIV Sinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Immune Enhancement Project (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 243A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-09

CONDITIONS: HIV Infections; Sinusitis
Keywords: AIDS-Related Opportunistic Infections; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Sinusitis; Ephedrine; Acupuncture Therapy; Drugs, Chinese Herbal; Medicine, Chinese Traditional; Drug Combinations; Antibiotics, Combined; Amoxicillin-Potassium Clavulanate Combination
MeSH Terms: conditions — HIV Infections; Sinusitis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Clavulanic Acid; Pseudoephedrine; Amoxicillin

INTERVENTIONS:
Drug: Clavulanate potassium
Drug: Pseudoephedrine hydrochloride
Drug: Amoxicillin trihydrate

SUMMARY:
To compare Traditional Chinese Medicine versus standard antibiotic therapy consisting of pseudoephedrine ( Sudafed ) plus amoxicillin / clavulanate potassium combination ( Augmentin ) in reducing symptoms and recurrence of acute HIV-related sinusitis.

Chronic sinusitis in HIV-infected individuals is a recurrent and persistent infection with potentially serious complications: it can exacerbate pulmonary disease, cause recurrences of life-threatening sepsis, and progress to central nervous system involvement. Symptoms of sinusitis in HIV patients are often refractory to aggressive Western medical management, and antibiotic intolerance can occur. Traditional Chinese Medicine consisting of acupuncture and herbal treatment may provide a low-risk, low-cost alternative to conventional antibiotic therapy.

DETAILED DESCRIPTION:
Chronic sinusitis in HIV-infected individuals is a recurrent and persistent infection with potentially serious complications: it can exacerbate pulmonary disease, cause recurrences of life-threatening sepsis, and progress to central nervous system involvement. Symptoms of sinusitis in HIV patients are often refractory to aggressive Western medical management, and antibiotic intolerance can occur. Traditional Chinese Medicine consisting of acupuncture and herbal treatment may provide a low-risk, low-cost alternative to conventional antibiotic therapy.

Patients are randomized to receive either Traditional Chinese Medicine (acupuncture and herbal treatment) or conventional antibiotic therapy (Sudafed and Augmentin). Treatment continues for 8 weeks, followed by a 4 week washout, with final follow-up at week 12. Patients must undergo endoscopic nasal exam and CT scan of paranasal sinus prior to study entry and at week 12.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiviral medication.

Patients must have:

* HIV infection.
* CD4 count >= 50 cells/mm3.
* Recurrent sinusitis.
* No active opportunistic infection.
* No disease progression.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active infection with fever > 102 F.
* Neurological symptoms such as epidural abscess, subdural hematoma, meningitis, and dementia.
* Malignant neoplasm of nasal passages.
* Not expected to remain clinically stable for the next 6 months.
* Inability to comply with protocol requirements.
* Malabsorption or inability to take oral medication.
* Concurrent participation on another study where antibiotics will be used.

Concurrent Medication:

Excluded:

* Antibiotics other than Septra.

Concurrent Treatment:

Excluded:

* Chinese herbal medicine or acupuncture unless on that study arm.
* Surgical intervention that has abated symptoms.

Patients with the following prior condition are excluded:

History of allergic reaction to the study antibiotics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (1):
- Immune Enhancement Project, San Francisco, California, United States